CLINICAL TRIAL: NCT02902939
Title: Myeloid-Derived Supressor Cells in Uncomplicated vs Complicated Patients After Cardiac Surgery
Brief Title: Myeloid-Derived Supressor Cells in Cardiac Surgery Patients
Acronym: MyDeCCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Evgeny Grigoryev, professor, the deputy director for scientific and clinical affairs, senior research specialist, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20161101
Record Dates: First submitted 2016-09-04; First posted 2016-09-16 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Insufficiency; Cardiac, Complicating Surgery; Systemic Inflammatory Response Syndrome
Keywords: Immune Suppression, Inflammatory Response, Cardiac Surgery
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncomplicated cardiac surgery patients (No Intervention): Patients after scheduled cardiac surgery procedures
- Complicated cardiac surgery patients (Active Comparator): MECC systems Cytokines modulation by CytoSorb and PMMA membranes
  Interventions: Device: minimal extracorporeal circulation (MEC); Procedure: The cytokines modulations

INTERVENTIONS:
Device: minimal extracorporeal circulation (MEC) — We should use the modification of extracorporeal circulation to reduce the systemic inflammatory response due to excessive haemodilution, allogenic blood transfusion.
  Arms: Complicated cardiac surgery patients
Procedure: The cytokines modulations — We should use the modification of cytokines by CytoSorb devices and cytokines removal by PMMA membranes during extracorporeal circulation in patients with risk factors of complications (long duration of extracorporeal circulation, re-do procedures and other)
  Other Names: CytoSorb devices,
  Arms: Complicated cardiac surgery patients

SUMMARY:
Pro- and anti-inflammatory response during the formation of the critical state develops at the same time. Because of its balanced or unbalanced systemic inflammation can be either aborted or able to lead to multiple organ failure. With regard to sepsis, systemic inflammatory response characteristics are well understood, is not achieved in respect of the "sterile" inflammation.

Extracorporeal circulation is a clinical model of systemic inflammatory response due to non-physiological activation of tissue factor in the extracorporeal perfusion, the use of non-pulsatile circulation mode, intentional / unintentional hypothermia, bacterial translocation from the gastrointestinal tract and perfusion deficit.

We have proved that the monocytes demonstrate suppressor function, which can be a predictor of complications from cardiac surgery patients.

The most important component of the formation of multiple organ failure (MOF) in critically ill patients is immunosuppression.

During the study of experimental and clinical tumor growth process scientists has provided a new population of immature myeloid cells (myeloid suppressor cells or suppressor cells of myeloid origin, MDSC). Most of the works have been devoted to the role of MDSC in the development of tumors, where it has been clearly shown that this cell population has an undoubted effect of immune suppression. However, recent studies show that the role of MDSC is not limited to cancer process, but extends to chronic or acute inflammation.

The aim of this study is to determine the role of MDSC in the development of immune suppression and complications after heart surgery carried out under cardiopulmonary bypass.

DETAILED DESCRIPTION:
The use of MEC systems can be useful to prevent the MDSC activation after cardiac surgery.

The procedures to modulate the cytokines concentration can be useful to prevent the MDSC activation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. the patients with ischemia heart disease and/or valvular heart disease,
2. signed inform consent,
3. CABG and/or valve replacement/plastic procedures.

Exclusion Criteria:

1) congenital heart disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
MOF-free days | 28 day

SECONDARY OUTCOMES:
ICU length of stay | 28 day
the incidents of infection complications | 28 day

CONTACTS AND LOCATIONS:
Locations (1):
- Georgy Plotnikov, Kemerovo, Russia

IPD SHARING:
Plan to Share IPD: No